CLINICAL TRIAL: NCT02873585
Title: Clinical Evaluation and Patient Experience of a Stationary Intraoral Tomosynthesis (s-IOT) Unit Using a Carbon Nanotube X-ray Source Array
Brief Title: Conventional Bite Wing Radiography Versus Stationary Intraoral Tomosynthesis, a Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: XinVivo, Inc. (Industry); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-0194
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stationary intraoral tomosynthesis (Experimental): Stationary intraoral tomosynthesis after standard conventional bitewing radiography
  Interventions: Device: Stationary intraoral tomosynthesis; Device: Standard conventional bitewing radiography

INTERVENTIONS:
Device: Stationary intraoral tomosynthesis — Bitewing radiographs using a stationary intraoral tomosynthesis unit
  Other Names: Dental tomosynthesis
Device: Standard conventional bitewing radiography — Bitewing radiographs using a stationary intraoral tomosynthesis unit will be performed after standard bitewing radiography

SUMMARY:
A comparison of caries detection rates between conventional intraoral bitewing radiography and a stationary intraoral digital tomosynthesis (s-IOT) using a carbon nanotube X-ray source array. The secondary objective is to assess participants experience with the s-IOT device.

DETAILED DESCRIPTION:
The primary purpose of this study is to compare caries detection rates between conventional intraoral bitewing radiography and a stationary intraoral digital tomosynthesis (s-IOT) using a carbon nanotube X-ray source array. Patient experience with the s-IOT device will be assess using a short questionnaire.

Fifty adult patients who have been referred to the Section of Oral and Maxillofacial Radiology (OMR) at the University of North Carolina (UNC) School of Dentistry (SOD) for horizontal bitewing (BW) radiographs or a Full Mouth Series (FMX) with horizontal bitewing radiographs will be recruited for the study.

Participants will receive an experimental s-IOT bitewing radiograph on each side of their mouth and a visual exam to look for caries. Experienced observers will assess the presence or absence of caries using the two imaging modalities. The results of their analysis will be evaluated to determine statistical difference. Participants completed questionnaires will be tabulated and the data will be analyzed using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Scheduled for horizontal BW or Full (FMX) with horizontal BWs
* Patients who have in the right and left maxilla and mandible at least a canine and two posterior teeth that are in contact
* At least one proximal caries lesion in a surface of a posterior tooth (premolar or molar) that is in contact with another tooth. Lesion depth can be incipient (outer half enamel), moderate (inner half enamel) or advanced (outer half dentin) as determined by conventional BW radiography.
* At least one non-carious proximal surface of a posterior tooth (premolar or molar) that is in contact with another tooth.
* Patients should be able to provide informed consent

Exclusion Criteria:

* Institutionalized subject (prisoners, nursing home, etc.) (identified by medical record)
* Critically ill or mentally unstable patients (identified by medical record)
* Patients with no radiographic caries of the posterior teeth as determined by conventional BW radiographs
* Patients with only severe caries lesions as determined by conventional BW radiographs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Broome, DDS, Principal Investigator — UNC-School of Dentistry
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Tooth surface
Period: Overall Study
Arm/Group | Stationary Intraoral Tomosynthesis
Started | 32; 217 Tooth surface
Completed | 32; 217 Tooth surface
Not Completed | 0; 0 Tooth surface

BASELINE CHARACTERISTICS:
Units Other Than Participants: Tooth Surfaces
Arm/Group | Stationary Intraoral Tomosynthesis
Number analyzed (Participants) | 32
Number analyzed (Tooth Surfaces) | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: ROC Using the Area Under the Curve (AUC)
Description: This prospective study is to compare the diagnostic performance (accuracy) of a stationary intraoral tomosynthesis device using a Carbon Nanotube X-ray source array and a conventional intraoral X-ray device in the diagnosis of interproximal caries. receiver operating characteristic (ROC) analysis will be used to compare the areas under the curve (AUC).
Time Frame: Within 7 months of last participants imaging
Measure: Mean (Standard Deviation); unit: probability
Units Other Than Participants: Tooth Surfaces
Groups:
- Standard Conventional Bitewing Radiography: Bitewing radiographs using a standard two-dimensional bitewing radiography
Arm/Group | Standard Conventional Bitewing Radiography | Stationary Intraoral Tomosynthesis
Number analyzed (Participants) | 32 | 32
Number analyzed (Tooth Surfaces) | 217 | 217
probability | 0.5427 (0.0473) | 0.5173 (0.0200)

2. Primary Outcome: Proportion of Healthy Tooth Surfaces
Description: Specificity reflects the ability of the system to correctly identify healthy tooth surfaces expressed as a proportion.
Time Frame: Within 7 months of last participants imaging
Measure: Mean (Standard Deviation); unit: proportion of tooth surfaces
Units Other Than Participants: tooth surfaces
Arm/Group | Standard Conventional Bitewing Radiography | Stationary Intraoral Tomosynthesis
Number analyzed (Participants) | 32 | 32
Number analyzed (tooth surfaces) | 217 | 217
proportion of tooth surfaces | 0.7308 (0.099) | 0.7657 (0.045)

3. Primary Outcome: Proportion of Carious Tooth Surfaces
Description: Sensitivity reflects the ability of the system to correctly identify carious tooth surfaces expressed as a proportion.
Time Frame: Within 7 months of last participants imaging
Measure: Mean (Standard Deviation); unit: proportion of carious tooth surfaces
Units Other Than Participants: tooth surfaces
Arm/Group | Standard Conventional Bitewing Radiography | Stationary Intraoral Tomosynthesis
Number analyzed (Participants) | 32 | 32
Number analyzed (tooth surfaces) | 217 | 217
proportion of carious tooth surfaces | 0.3601 (0.1006) | 0.2768 (0.0401)

4. Secondary Outcome: Number of Participants With a Positive Experience
Description: Questionnaire used a five point Likert scale for evaluating participants' comfort with the experimental tomosynthesis unit (s-IOT) when compared to the standard intraoral unit used for bitewing radiography. Survey was distributed immediately after the examination using the experimental tomosynthesis unit. A score of 1 reflects "strongly disagree" and a score of 5 reflects "strongly disagree." A "positive experience" was defined as a score greater than 3.
Time Frame: During a single 2-hour visit
Population: Responses reported for all that were received
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Conventional Bitewing Radiography | Stationary Intraoral Tomosynthesis
Number analyzed (Participants) | 32 | 32
Participants
  Equally Comfortable | 13 | 19
  More Comfortable: number analyzed (Participants) | 26 | 26
  More Comfortable | 8 | 18
  Requires More Time: number analyzed (Participants) | 31 | 31
  Requires More Time | 6 | 25
  Equally Easy to Perform | 16 | 16
  More Difficult to Perform | 14 | 18
  Noticeably Different | 18 | 14
  Recommended Without Reservation | 27 | 5
  Reported No Issues with Either System: number analyzed (Participants) | 28 | 28
  Reported No Issues with Either System | 18 | 10

5. Secondary Outcome: Overall Investigator Confidence Survey
Description: The investigators were to complete a brief survey regarding the overall confidence in diagnosis, time, and the number of required radiographic re-takes.
Time Frame: During a single 2-hour visit
Population: This survey tool was not developed or executed; therefore, these data were not collected.
Arm/Group | Stationary Intraoral Tomosynthesis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: During a single 2-hour visit.
Arm/Group | Standard Conventional Bitewing Radiography | Stationary Intraoral Tomosynthesis
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT02873585/Prot_SAP_000.pdf